CLINICAL TRIAL: NCT01803568
Title: Skeletal Muscles, Myokines and Glucose Metabolism
Brief Title: Skeletal Muscles, Myokines and Glucose Metabolism MYOGLU
Acronym: MyoGlu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Kåre Inge Birkeland, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011/882
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Hyperglycemia; Normoglycemia; Myokine
Keywords: Myokine; Insulin sensitivity; Exercise; Skeletal muscle
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise in normoglycaemic individuals (Experimental)
  Interventions: Other: Exercise
- Exercise in hyperglycaemic individuals (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 12 weeks of exercise; 4 times pr week

SUMMARY:
Normal glucose uptake and metabolism in skeletal muscles are essential to keep blood glucose within normal range and hence, insulin resistance (possibly mediated by inflammatory processes) in skeletal muscle is a major pathogenic factor in type 2 diabetes. Physical activity seems to be of essential importance in the prevention and treatment of type 2 diabetes. Myokines are proteins secreted from skeletal muscle that can execute important biological functions locally in the muscle (paracrine) or in other organs like the brain, heart and pancreas (endocrine). Evidence suggest that several interleukines and other cytokines are secreted by skeletal muscles. In the present project, the investigators will explore the relation between secreted myokines from muscle cells, insulin resistance and glucose metabolism before and after 12 weeks of exercise intervention. Subjects with normal as well as impaired glucose metabolism will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 40-65 years
* Nordic ethnicity
* Non-smoker

  1. Either (participants with impaired glucose metabolism): Body Mass Index (BMI) 27-32 kg/m2 and abnormal glucose metabolism, defined as:

     i. impaired fasting glucose (FPG ≥ 5.6 mmol/L) ii. impaired glucose tolerance (2 h PG ≥7.8 mmol/L) iii. type 2 diabetes (no medication, HbA1c ≤7.5%)
  2. Or (controls): BMI 19-25 kg/m2 and normal glucose metabolism and no first degree relatives with type 2 diabetes.

Exclusion Criteria:

1. Subjects having type 1 diabetes or medically treated type 2 diabetes.
2. Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 90 mmHg at screening
3. Significant hematological or renal disease or chronic renal impairment, GFR< 50 ml/min.
4. Significant liver disease or ALAT >3x UNL.
5. Chronic inflammatory disease in active phase or long-term use of corticosteroids last 3 months.
6. Use of anti-diabetic agents, lipid lowering drugs, antihypertensive medication, ASA or any other drug not deemed suitable by the study physician.
7. Mental condition (psychiatric or organic cerebral disease), drug or alcohol abuse rendering the subject unable to understand the nature, scope and possible consequences of the study.
8. BMI outside inclusion criteria.
9. Smoker
10. Any medical or other condition that in the judgment of the investigator would jeopardize the subject's safety or evaluation of the intervention for efficacy and safety
11. Exercising regularly (>1 times pr week)

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in gene expression changes in skeletal and adipose tissue | Baseline and after 12 weeks, and before, 0 hr and 2 hours after acute exercise
Changes from baseline in plasma/serum levels of selected proteins | Baseline and after 12 weeks, and before, 0 hr and 2 hour

SECONDARY OUTCOMES:
Change from baseline in insulin sensitivity | Before and after 12 weeks of exercise
  Insulin sensitivity will be measured using the euglycaemic hyperinsulinaemic clamp technique.
Changes in baseline from maximal oxygen uptake VO2 max | Before and after 12 weeks
Changes from baseline in muscle strength | Before and after 12 weeks
Changes from baseline in body composition | Before and after 12 weeks
  Body composition will be estimated with whole body MRI.
Changes from baseline in heart frequency | Before and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kåre I Birkeland, MD PhD, Principal Investigator — Oslo University Hospital; Christian A Drevon, MD PhD, Study Chair — University of Oslo

REFERENCES:
- [Derived] Lee-Odegard S, Austin Argentieri M, Norheim F, Drevon CA, Birkeland KI. Reversal of proteomic aging with exercise-results from the UK biobank and a 12-week intervention study. NPJ Aging. 2025 Dec 26. doi: 10.1038/s41514-025-00318-w. Online ahead of print. PMID 41449222
- [Derived] Lee-Odegard S, Hjorth M, Olsen T, Moen GH, Daubney E, Evans DM, Hevener AL, Lusis AJ, Zhou M, Seldin MM, Allayee H, Hilser J, Viken JK, Gulseth H, Norheim F, Drevon CA, Birkeland KI. Serum proteomic profiling of physical activity reveals CD300LG as a novel exerkine with a potential causal link to glucose homeostasis. Elife. 2024 Aug 27;13:RP96535. doi: 10.7554/eLife.96535. PMID 39190027
- [Derived] Doncheva AI, Romero S, Ramirez-Garrastacho M, Lee S, Kolnes KJ, Tangen DS, Olsen T, Drevon CA, Llorente A, Dalen KT, Hjorth M. Extracellular vesicles and microRNAs are altered in response to exercise, insulin sensitivity and overweight. Acta Physiol (Oxf). 2022 Dec;236(4):e13862. doi: 10.1111/apha.13862. Epub 2022 Aug 10. PMID 36377504
- [Derived] Moore TM, Zhou Z, Cohn W, Norheim F, Lin AJ, Kalajian N, Strumwasser AR, Cory K, Whitney K, Ho T, Ho T, Lee JL, Rucker DH, Shirihai O, van der Bliek AM, Whitelegge JP, Seldin MM, Lusis AJ, Lee S, Drevon CA, Mahata SK, Turcotte LP, Hevener AL. The impact of exercise on mitochondrial dynamics and the role of Drp1 in exercise performance and training adaptations in skeletal muscle. Mol Metab. 2019 Mar;21:51-67. doi: 10.1016/j.molmet.2018.11.012. Epub 2018 Dec 4. PMID 30591411
- [Derived] Lee S, Norheim F, Gulseth HL, Langleite TM, Aker A, Gundersen TE, Holen T, Birkeland KI, Drevon CA. Skeletal muscle phosphatidylcholine and phosphatidylethanolamine respond to exercise and influence insulin sensitivity in men. Sci Rep. 2018 Apr 25;8(1):6531. doi: 10.1038/s41598-018-24976-x. PMID 29695812
- [Derived] Sommer C, Lee S, Gulseth HL, Jensen J, Drevon CA, Birkeland KI. Soluble Leptin Receptor Predicts Insulin Sensitivity and Correlates With Upregulation of Metabolic Pathways in Men. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1024-1032. doi: 10.1210/jc.2017-02126. PMID 29300960
- [Derived] Lee S, Norheim F, Langleite TM, Noreng HJ, Storas TH, Afman LA, Frost G, Bell JD, Thomas EL, Kolnes KJ, Tangen DS, Stadheim HK, Gilfillan GD, Gulseth HL, Birkeland KI, Jensen J, Drevon CA, Holen T; NutriTech Consortium. Effect of energy restriction and physical exercise intervention on phenotypic flexibility as examined by transcriptomics analyses of mRNA from adipose tissue and whole body magnetic resonance imaging. Physiol Rep. 2016 Nov;4(21):e13019. doi: 10.14814/phy2.13019. PMID 27821717